CLINICAL TRIAL: NCT02672514
Title: Does Minimal Extracorporeal Circulation Improve Outcome in Diabetic Patients Undergoing Elective Coronary Bypass Grafting?
Brief Title: Does MiECC Improve Outcome in Diabetic Patients Undergoing Elective Coronary Bypass Grafting?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herzzentrum Coswig (Other)
Responsible Party: Principal Investigator, PD Dr. Hausmann, chief physician, Herzzentrum Coswig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rölig Studie
Record Dates: First submitted 2016-01-19; First posted 2016-02-03 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- MiECC (Active Comparator): Coronary artery bypass grafting is used with the help of cardiopulmonary bypass (CPB). The technique used in this arm based on the minimally invasive extracorporeal circulation system (MiECC). MiECC has been developed based on the concept of a closed total CPB circuit. The basic elements are a centrifugal pump, a membrane oxygenator and an arterial filter. The priming volume compared to CECC could be reduced. The complete circuit is heparin-coated for maximizing the biocompatibility.
  CPB was performed under normothermic conditions of 36°C. Retrograde autologous priming was performed for all patients with stable hemodynamic circulation.
  Interventions: Device: Minimally invasive extracorporeal circulation (MiECC)
- CECC (Active Comparator): Coronary artery bypass grafting is used with the help of cardiopulmonary bypass (CPB). The technique used in this arm based on the conventional extracorporeal circulation system (CECC). The CECC is an opened circulation system. The basic elements are a membrane oxygenator, a centrifugal pump, an open perfusion system containing the venous hard shell cardiotomy reservoir and the arterial line filter.
  CPB was performed under normothermic conditions of 36°C. Retrograde autologous priming was performed for all patients with stable hemodynamic circulation, leading to a reduction of the priming volume. The CECC flow was set as required in order to maintain a mean arterial pressure (MAP) between 50 and 75 mmHg.
  Interventions: Device: Conventional extracorporeal circulation (CECC)

INTERVENTIONS:
Device: Minimally invasive extracorporeal circulation (MiECC) — Minimally invasive extracorporeal circulation (MiECC) is an extracorporeal circulation systems used for cardiopulmonary bypass.
  Arms: MiECC
Device: Conventional extracorporeal circulation (CECC) — Conventional extracorporeal circulation (CECC) is an extracorporeal circulation system used for cardiopulmonary bypass.
  Arms: CECC

SUMMARY:
The aim of this study was to prospectively evaluate MECC compared with conventional extracorporeal circulation of diabetic patients undergoing elective coronary revascularization procedures. The investigators focused on the effects of extracorporeal circulation especially the renal function between both groups.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) is known having a negative influence referring to systemic inflammatory reaction after cardiac surgery which can cause acute kidney injury (AKI). Miniaturized extracorporeal circulation (MECC) attempts to reduce the adverse effects of conventional extracorporeal circulation bypass. Finally, AKI after CPB is a significant clinical problem that increasingly complicates the course of hospitalization and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus type 2
* isolated elective coronary revascularization

Exclusion Criteria:

* urgent or emergent Status
* Re-Operation
* preexisting reanimation
* preexisting renal transplantation
* chronic kidney insufficiency (GFR < 30 ml/min)
* renal cell carcinoma
* renal artery Stenosis
* heart valve disease (middle- and high-grade)
* endocarditis
* infections (HIV, Tbc and all types of Hepatitis)
* hepatic cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-02; Primary Completion 2012-04 (Actual); Study Completion 2015-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- MiECC: Coronary artery bypass grafting is used with the help of cardiopulmonary bypass (CPB). The technique used in this arm based on the minimally invasive extracorporeal circulation system (MiECC). MiECC has been developed based on the concept of a closed total CPB circuit. The basic elements are a centrifugal pump, a membrane oxygenator and an arterial filter. The priming volume compared to CECC could be reduced. The complete circuit is heparin-coated for maximizing the biocompatibility.
  CPB was performed under normothermic conditions of 36°C. Retrograde autologous priming was performed for all patients with stable hemodynamic circulation.
  Minimally invasive extracorporeal circulation (MiECC): Minimally invasive extracorporeal circulation (MiECC) is an extracorporeal circulation systems used for cardiopulmonary bypass.
- CECC: Coronary artery bypass grafting is used with the help of cardiopulmonary bypass (CPB). The technique used in this arm based on the conventional extracorporeal circulation system (CECC). The CECC is an opened circulation system. The basic elements are a membrane oxygenator, a centrifugal pump, an open perfusion system containing the venous hard shell cardiotomy reservoir and the arterial line filter.
  CPB was performed under normothermic conditions of 36°C. Retrograde autologous priming was performed for all patients with stable hemodynamic circulation, leading to a reduction of the priming volume. The CECC flow was set as required in order to maintain a mean arterial pressure (MAP) between 50 and 75 mmHg.
  Conventional extracorporeal circulation (CECC): Conventional extracorporeal circulation (CECC) is an extracorporeal circulation system used for cardiopulmonary bypass.
Period: Overall Study
Arm/Group | MiECC | CECC
Started | 53 | 51
Completed | 53 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group B: Coronary artery bypass grafting is used with the help of cardiopulmonary bypass (CPB). The technique used in this arm based on the minimally invasive extracorporeal circulation system (MiECC). MiECC has been developed based on the concept of a closed total CPB circuit. The basic elements are a centrifugal pump, a membrane oxygenator and an arterial filter. The priming volume compared to CECC could be reduced. The complete circuit is heparin-coated for maximizing the biocompatibility.
  CPB was performed under normothermic conditions of 36°C. Retrograde autologous priming was performed for all patients with stable hemodynamic circulation.
  Minimally invasive extracorporeal circulation (MiECC): Minimally invasive extracorporeal circulation (MiECC) is an extracorporeal circulation systems used for cardiopulmonary bypass.
- Group A: Coronary artery bypass grafting is used with the help of cardiopulmonary bypass (CPB). The technique used in this arm based on the conventional extracorporeal circulation system (CECC). The CECC is an opened circulation system. The basic elements are a membrane oxygenator, a centrifugal pump, an open perfusion system containing the venous hard shell cardiotomy reservoir and the arterial line filter.
  CPB was performed under normothermic conditions of 36°C. Retrograde autologous priming was performed for all patients with stable hemodynamic circulation, leading to a reduction of the priming volume. The CECC flow was set as required in order to maintain a mean arterial pressure (MAP) between 50 and 75 mmHg.
  Conventional extracorporeal circulation (CECC): Conventional extracorporeal circulation (CECC) is an extracorporeal circulation system used for cardiopulmonary bypass.
- Total: Total of all reporting groups
Arm/Group | Group B | Group A | Total
Number analyzed (Participants) | 53 | 51 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 27
  >=65 years | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.25 (8.95) | 67.98 (8.43) | 67.1 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: Acute Kidney Injury
Time Frame: within the first 30 days (plus or minus 3 days) after surgery
Measure: Number; unit: participants
Arm/Group | Group B | Group A
Number analyzed (Participants) | 53 | 51
participants
  direct after operation | 7 | 41
  1 hour after operation | 9 | 40
Statistical Analysis 1: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of serum Creatinine concentration. We test the null hypothesis that serum Creatinine was the same in both groups. The first blood samples from both groups were collected before cardiopulmonary bypass; Test type: Superiority or Other; p = 0.377, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of serum Creatinine concentration. We test the null hypothesis that serum Creatinine was the same in both groups. The blood samples were collected from both groups on arrival of intensive care unit; Test type: Superiority or Other; p = 0.051, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of serum Creatinine concentration. We test the null hypothesis that serum Creatinine was the same in both groups. The blood samples from both groups were collected 24 hours after Operation; Test type: Superiority or Other; p = 0.282, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of serum Creatinine concentration. We test the null hypothesis that serum Creatinine was the same in both groups. These blood samples were collected 48 hours after cardiopulmonary Bypass; Test type: Superiority or Other; p = 0.277, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of serum Creatinine concentration. We test the null hypothesis that serum Creatinine was the same in both groups. The blood samples were collected from both groups 72 hours after cardiopulmonary bypass; Test type: Superiority or Other; p = 0.308, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of serum Cystatin C concentration. We test the null hypothesis that serum Cystatin C was the same in both groups. The first blood samples were collected before cardiopulmonary bypass; Test type: Superiority or Other; p = 0.211, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of serum Cystatin C concentration. We test the null hypothesis that serum Cystatin C was the same in both groups. The blood samples were collected on arrival of intensive care unit; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of serum Cystatin C concentration. We test the null hypothesis that serum Cystatin C was the same in both groups. The blood samples were collected 24 hours after operation; Test type: Superiority or Other; p = 0.221, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of serum Cystatin C concentration. We test the null hypothesis that serum Cystatin C was the same in both groups. The blood samples were collected 48 hours after operation; Test type: Superiority or Other; p = 0.796, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of serum Cystatin C concentration. We test the null hypothesis that serum Cystatin C was the same in both groups. The blood samples were collected 72 hours after operation; Test type: Superiority or Other; p = 0.463, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of the postoperative NGAL levels in plasma. We test the null hypothesis that the NGAL level was the same in both groups. The first blood samples were collected before cardiopulmonary bypass; Test type: Superiority or Other; p = 0.118, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of the postoperative NGAL levels in plasma. We test the null hypothesis that the NGAL level was the same in both groups. The blood samples were collected on arrival of intensive care unit; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of the postoperative NGAL levels in plasma. We test the null hypothesis that the NGAL level was the same in both groups. The blood samples were collected one hour after cardiopulmonary bypass; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of the postoperative NGAL levels in plasma. We test the null hypothesis that the NGAL level was the same in both groups. The blood samples were collected four hours after cardiopulmonary bypass; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Group B vs Group A; The early diagnosis of AKI currently depends on the detection of reduced kidney function by the rise of the postoperative NGAL levels in plasma. We test the null hypothesis that the NGAL level was the same in both groups. The blood samples were collected 48 hours after cardiopulmonary bypass; Test type: Superiority or Other; p = 0.171, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | MiECC | CECC
Serious Adverse Events (participants affected / at risk) | 12/53 | 7/51
Other Adverse Events (participants affected / at risk) | 0/53 | 1/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MiECC (N=53) | CECC (N=51)
dialysis (Blood and lymphatic system disorders) | 1 | 2
cardiogenic shock (Cardiac disorders) | 1 | 1
perioperative myocardial infarction (Cardiac disorders) | 1 | 0
pericardial effusion (Cardiac disorders) | 2 | 0
reanimation (General disorders) | 1 | 1
re-operation (Surgical and medical procedures) | 3 | 2
re-PTCA (Surgical and medical procedures) | 3 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MiECC (N=53) | CECC (N=51)
use of IABP (Surgical and medical procedures) | 0 | 1

LIMITATIONS AND CAVEATS:
only a single-Center study; a small number of study participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No